CLINICAL TRIAL: NCT07053345
Title: An Interventional, Open-label, Single Arm, Multicenter Study to Evaluate the Efficacy and Safety of Esketamine Nasal Spray in Korean Participants With Treatment-Resistant Depression(TRD)
Brief Title: A Study of Esketamine Nasal Spray in Korean Participants With Treatment-resistant Depression
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Janssen Korea, Ltd., Korea (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 54135419TRD4017; 54135419TRD4017 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2025-06-27; First posted 2025-07-08 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Depressive Disorder, Treatment-Resistant
MeSH Terms: conditions — Depressive Disorder, Treatment-Resistant | interventions — Esketamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Esketamine Nasal Spray (Experimental): Participants will self-administer one esketamine (flexibly dosed; 56 or 84 milligrams [mg]) nasal spray into each nostril (that is, a total of 2 sprays using 1 intranasal device) twice a week for 4 weeks. For 84 mg, sprays to each nostril will be delivered in rapid succession at 3 different time points (3 devices total). 56 mg will have 2 devices.
  Interventions: Drug: Esketamine 56 mg; Drug: Esketamine 84 mg

INTERVENTIONS:
Drug: Esketamine 56 mg — Participants will self-administer 56 mg of esketamine as intranasal spray into each nostril.
  Other Names: JNJ-54135419
Drug: Esketamine 84 mg — Participants will self-administer 84 mg of esketamine as intranasal spray into each nostril.
  Other Names: JNJ-54135419

SUMMARY:
The purpose of this study is to evaluate how well esketamine nasal spray works in improving depressive symptoms in participants with treatment resistant depression (TRD). This will be assessed by the change from baseline in the Hamilton depression rating scale (HAM-D; 17-item) total score from Day 1 (baseline) to the end of the 4-week treatment phase (Day 28).

ELIGIBILITY:
Inclusion Criteria:

* Must have a confirmed diagnosis of major depressive disorder (MDD) according to the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition at the time of enrollment, without psychotic features, based on clinical assessment, and confirmed by mini international neuropsychiatric interview (MINI)
* Must have a Hamilton depression rating scale (HAM-D; 17-item) total score greater than or equal to (>=) 22 at screening and Day 1
* Participants must have had non-response (less than or equal to [<=] 25 percent [%] improvement of symptoms) to >= 2 oral antidepressant treatments in the current moderate to severe episode of depression after having been given at an adequate dosage for an adequate duration of at least 6 weeks
* At baseline (Day 1), the investigator will evaluate any changes in the participant's signs/symptoms of depression since the screening assessment and confirm that the inclusion criteria for the current antidepressant (AD) treatment are still met (that is, nonresponse and minimal clinical improvement)
* A female participant of childbearing potential must have a negative serum pregnancy test at screening and urine prior to the first dose of study intervention on Day 1

Exclusion Criteria:

* Participants with hyperthyroidism that has not been sufficiently treated
* History of malignancy within 5 years of enrollment before screening
* Known allergies, hypersensitivity, or intolerance to esketamine/ketamine or its excipients
* Received an investigational intervention or used an invasive investigational medical device within 60 days before the planned first dose of study intervention or first data collection time point
* Currently enrolled in an investigational study that involves treatments for MDD or may otherwise be expected to impact mood

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 47 (Estimated)
Dates: Start 2025-06-09 (Actual); Primary Completion 2027-06-25 (Estimated); Study Completion 2027-06-25 (Estimated)

PRIMARY OUTCOMES:
Change From Baseline to Day 28 in Hamilton Depression Rating Scale (HAM-D) Total Score | Baseline up to Day 28
  The HAM-D contains 17 items pertaining to symptoms of depression experienced over the past week. The questions cover core symptoms of depression as well as appetite and sleep (3 items). Items are scored on a likert scale of 0-4 or 0-2 depending on the item with a possible range of 0-52, with higher scores indicating greater severity of depressive symptoms.

SECONDARY OUTCOMES:
Change From Baseline Over Time for HAM-D Total Score | Baseline up to Week 4
  The HAM-D contains 17 items pertaining to symptoms of depression experienced over the past week. The questions cover core symptoms of depression as well as appetite and sleep (3 items). Items are scored on a likert scale of 0-4 or 0-2 depending on the item with a possible range of 0-52, with higher scores indicating greater severity of depressive symptoms.
Change From Baseline Over Time for Patient Health Questionnaire 9-item (PHQ-9) Total Score | Baseline up to Week 4
  The PHQ-9 is a validated 9-item, patient-reported outcomes (PRO) measure to assess depressive symptoms. The scale scores each of the 9 symptom domains of the diagnostic and statistical manual of mental disorders, fifth edition (DSM-5) major depressive disorder (MDD) criteria and it has been used both as a screening tool and a measure of response to treatment for depression. Each item is rated on a 4-point scale (0=not at all, 1=several days, 2=more than half the days, and 3=nearly every day). The participant's item responses are summed to provide a total score (range of 0 to 27), with higher scores indicating greater severity of depressive symptoms.
Percentage of Participants With Response Based on HAM-D Total Score Over Time | Up to Week 4
  Percentage of participants with response based on HAM-D total score over time will be reported. The HAM-D contains 17 items pertaining to symptoms of depression experienced over the past week. The questions cover core symptoms of depression as well as appetite and sleep (3 items). Items are scored on a likert scale of 0-4 or 0-2 depending on the item with a possible range of 0-52, with higher scores indicating greater severity of depressive symptoms.
Percentage of Participants With Response Based on PHQ-9 Total Score Over Time | Up to Week 4
  Percentage of participants with response based on PHQ-9 total score over time will be reported. The PHQ-9 is a validated 9-item, PRO measure to assess depressive symptoms. The scale scores each of the 9 symptom domains of the DSM-5 MDD criteria and it has been used both as a screening tool and a measure of response to treatment for depression. Each item is rated on a 4-point scale (0=not at all, 1=several days, 2=more than half the days, and 3=nearly every day). The participant's item responses are summed to provide a total score (range of 0 to 27), with higher scores indicating greater severity of depressive symptoms.
Percentage of Participants With Remission Based on HAM-D Total Score Over Time | Up to Week 4
  Percentage of participants with remission based on HAM-D total score over time will be reported. The HAM-D contains 17 items pertaining to symptoms of depression experienced over the past week. The questions cover core symptoms of depression as well as appetite and sleep (3 items). Items are scored on a likert scale of 0-4 or 0-2 depending on the item with a possible range of 0-52, with higher scores indicating greater severity of depressive symptoms.
Percentage of Participants With Remission Based on PHQ-9 Total Score Over Time | Up to Week 4
  Percentage of participants with remission based on PHQ-9 total score over time will be reported. The PHQ-9 is a validated 9-item, PRO measure to assess depressive symptoms. The scale scores each of the 9 symptom domains of the DSM-5 MDD criteria and it has been used both as a screening tool and a measure of response to treatment for depression. Each item is rated on a 4-point scale (0=not at all, 1=several days, 2=more than half the days, and 3=nearly every day). The participant's item responses are summed to provide a total score (range of 0 to 27), with higher scores indicating greater severity of depressive symptoms.
Percentage of Participants With Clinically Meaningful Improvement Based on HAM-D Total Score Over Time | Up to Week 4
  Percentage of participants with clinically meaningful improvement based on HAM-D total score over time will be reported. The HAM-D contains 17 items pertaining to symptoms of depression experienced over the past week. The questions cover core symptoms of depression as well as appetite and sleep (3 items). Items are scored on a likert scale of 0-4 or 0-2 depending on the item with a possible range of 0-52, with higher scores indicating greater severity of depressive symptoms.
Percentage of Participants With Clinically Meaningful Improvement Based on PHQ-9 Total Score Over Time | Up to Week 4
  Percentage of participants with clinically meaningful improvement based on total score PHQ-9 total score over time will be reported. The PHQ-9 is a validated 9-item, PRO measure to assess depressive symptoms. The scale scores each of the 9 symptom domains of the DSM-5 MDD criteria and it has been used both as a screening tool and a measure of response to treatment for depression. Each item is rated on a 4-point scale (0=not at all, 1=several days, 2=more than half the days, and 3=nearly every day). The participant's item responses are summed to provide a total score (range of 0 to 27), with higher scores indicating greater severity of depressive symptoms.
Change From Baseline Over Time for Clinical Global Impression-Severity (CGI-S) Score | Baseline up to Week 4
  The CGI-S is a clinician-rated scales that measure illness severity. The CGI has proved to be a robust measure of efficacy in many clinical drug trials and is easy and quick to administer. The CGI-S is rated on a 7-point scale, with the severity of illness scale using a range of responses from 1 (normal) through to 7 (among the most severely ill participants).

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Korea, Ltd., Korea Clinical Trial, Study Director — Janssen Korea, Ltd., Korea
Locations (6):
- South Korea (6):
  - Cha Ilsan Medical Center, Goyang Si Gyeonggi Do
  - Wonkwang University Hospital, Iksan
  - Kyung Hee University Medical Center, Seoul
  - Kangbuk Samsung Hospital, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of Johnson & Johnson Innovative Medicine is available at innovativemedicine.jnj.com/our-innovation/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://innovativemedicine.jnj.com/our-innovation/clinical-trials/transparency